CLINICAL TRIAL: NCT05072418
Title: The Influence of Visual Information on Postural Control Among Children with and Without Dyslexia
Brief Title: Postural Control Among Children with and Without Dyslexia
Status: Completed | Type: Observational
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: A-BR-109-041
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Child Development Disorder
Keywords: child with dyslexia, postural sway; visual perception
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Children with dyslexia
  Interventions: Behavioral: Eye-opened and Eye-closed
- Non-dyslexic children
  Interventions: Behavioral: Eye-opened and Eye-closed

INTERVENTIONS:
Behavioral: Eye-opened and Eye-closed — The participants were instructed to perform six 60-second trials (2 conditions × 3 trials) of maintaining an upright stance on a force plate (Kistler Type 9260A, Switzerland) under the eyes open (EO) and eyes closed (EC) conditions. The order of EO and EC was alternated for each participant, and half of the subjects began with the EO (or EC) condition. For both conditions, the participants stood with their feet 1 cm apart on a force plate and their arms relaxed comfortably at their sides.

SUMMARY:
As Chinese-speaking children with dyslexia typically have different cerebellar sign behavior from non-Chinese-speaking counterparts, this study compared the effect of visual occlusion on the static balance between dyslexic and non-dyslexic children using the Chinese language.

ELIGIBILITY:
Inclusion Criteria:

* 1.Normal IQ(>85, WISC-III)
* 2.Children with dyslexia assessed by standard tools, performed by psychological-teachers of special education

Exclusion Criteria:

* 1.Attention deficit hyperactivity disorder(ADHD)
* 2.Neurological or psychiatric abnormalities
* 3.Developmental coordination disorder(DCD)

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The participants will be 80 Chinese-speaking children between 8 and 12 years of age recruited from elementary schools in Taiwan. Half of the participants will be formally identified as dyslexia by specialists in the field of special education (Table 1), based on formal psycho-educational assessments (Chinese Character Recognition Test (Huang, 2001), Chinese reading diagnostic evaluation, and Wechsler Intelligence Scale for Children 4th Edition-Chinese version.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-12-26 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Postural sway analysis | through study completion, an average of 1 year
  Root mean squared sway amplitude and sample entropy along the AP and ML axes

SECONDARY OUTCOMES:
Stabilogram diffusion analysis of central of pressure | through study completion, an average of 1 year
  Trajectories of central of pressure will be analyzed with stabilogram diffusion analysis to reveal behavior mechanisms for practice-related variations in feedback and feedforward process for error corrections

CONTACTS AND LOCATIONS:
Locations (1):
- National Chen Kong University Hospital, Tainan, Taiwan